CLINICAL TRIAL: NCT07147569
Title: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis Post-Marketing Surveillance
Brief Title: TAMBE Japan Post-Marketing Surveillance
Status: Not yet recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 25-02
Record Dates: First submitted 2025-08-19; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Pararenal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TAMBE
  Interventions: Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis — The target patients are those who were attempted to implant the AC during the enrollment period of this surveillance. Patients will also be targeted even if all components of the TAMBE device (devices that can be used in combination with AC specified in IFU) were not used, or if a device other than the component of the TAMBE device was used.

SUMMARY:
To evaluate the safety and efficacy of multi component system (TAMBE device) including GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (Aortic Component; AC) under post-marketing use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were attempted to implant the AC
* Thoracoabdominal aortic aneurysm
* Pararenal abdominal aortic aneurysm

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target patients are those who were attempted to implant the AC during the enrollment period of this surveillance. Patients will also be targeted even if all components of the TAMBE device (devices that can be used in combination with AC specified in IFU) were not used, or if a device other than the component of the TAMBE device was used.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2034-02-28 (Estimated); Study Completion 2034-02-28 (Estimated)

PRIMARY OUTCOMES:
Technical Success | From the initial incision or puncture of the access vessel for the implantation procedure to the closure of the access vessel
  Calculate the rate of achievement of technical success at the index procedure. The technical success is defined as follows.
  [Technical success]
  All of the following qualifying criteria are met:
  * Successful access to the access vessels
  * Successful delivery and deployment of AC and all stent grafts used in combination with AC to its intended location
  * Successful side branch delivery catheterization and placement of all stent grafts used in the side branch area to its intended location
  * Absence of type I or type III endoleaks at final completion image evaluation
  * Patency of AC and all stent grafts used in combination with AC at final completion image evaluation
  * Absence of open surgical repair conversion or mortality
Clinical Success | 12 Months
  The achievement rate of clinical success will be calculated. The clinical success is defined as follows.
  [Clinical Success]
  * Achievement of technical success
  * Absence of the events listed below from the time of the index procedure to 12 months after the index procedure
    1. Death from the index procedure
    2. Death from reintervention
    3. Death from aorta-related causes
    4. Persistent type I or type III endoleaks
    5. Lesion enlargement >5 mm
    6. Device migration >10 mm
    7. Failure due to device integrity issues
    8. Lesion rupture
    9. Conversion to open surgical repair
    10. Permanent paraplegia
    11. Disabling stroke
    12. New-onset dialysis
Results related to abdominal branch vessels | 60 Months
  Calculate the incidence of the following events related to abdominal branch vessels (celiac artery, superior mesenteric artery, left/ right renal arteries) or AC and stent grafts used in combination with AC for visceral branch vessels.
  * Primary Patency
  * Primary Assisted Patency
  * Secondary Patency
  * Occlusion
  * Stenosis
  * Kink
  * Target vessel instability
  * Intraprocedural Complications
Major Adverse Events (MAEs) | 60 Months
  The incidence of any of following events is calculated.
  * All-cause mortality
  * Myocardial infarction resulting in death, cardiac arrest, or cardiopulmonary resuscitation
  * Respiratory failure requiring prolonged (> 24 hours) mechanical ventilation or reintubation
  * Renal function decline characterized by one or more of the following:
    1. > 50% reduction in pre-treatment Estimated Glomerular Filtration Rate (eGFR)
    2. New-onset dialysis
  * Bowel ischemia requiring surgical resection or not resolving with medical therapy
  * Permanent paraplegia
  * Major stroke (Any fatal or disabling stroke).
Thirty-Day Mortality | 30 Days
  Calculate thirty-day mortality. Thirty-day mortality is defined as follows.
  [Thirty-Day Mortality]
  Any death that occurs at the index procedure, within the index procedure hospital stay, or within the first 30 days post-index procedure.
Lesion-Related Mortality | 30 Days
  Calculate lesion-related mortality. Lesion-related mortality is defined as follows.
  [Lesion-related mortality]
  Any death that occurs within the first 30 days, any death that results from lesion rupture, aorta-related adverse events (e.g., infection, occlusion, dissection, hematoma), or adverse events related to a secondary intervention.
Reintervention | 60 Months
  Calculate the incidence of reintervention. Reintervention will be classified as "major" or "minor". Reintervention and its classifications are defined as follows.
  [Reintervention]
  Any procedure after the index procedure on the AC and stent grafts used in combination with AC.
  [Major Reintervention]
  Deployment the stent graft for proximal or distal side, removal of AC and stent grafts used in combination with AC, use of thrombectomy or thrombolysis, and surgical procedure.
  [Minor Reintervention]
  Treatment other than major reintervention that falls under any of the following categories
  * Endovascular procedures (percutaneous transluminal angioplasty, atherectomy, stenting)
  * Interventions to treat branch vessel stenosis
  * Interventions to treat type II endoleaks or branch-related endoleaks.

IPD SHARING:
Plan to Share IPD: No